CLINICAL TRIAL: NCT01484119
Title: Multi-center, Double-blind, Double-dummy, Randomized, Placebo-controlled, Active-reference, Parallel-group Study to Evaluate the Efficacy, Safety, and Tolerability of ACT-129968 in Adolescent, Adult & Elderly Patients With Seasonal Allergic Rhinitis
Brief Title: Efficacy, Safety, and Tolerability Study of ACT-129968 in Patients With Seasonal Allergic Rhinitis
Acronym: SAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-060B307
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — 2-(2-(1-naphthoyl)-8-fluoro-3,4-dihydro-1H-pyrido(4,3-b)indol-5(2H)-yl)acetic acid; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational Drug (Active Comparator): ACT-129968
  Interventions: Drug: ACT-129968
- Comparative Drug (Placebo Comparator): matching placebo tablets and capsules
  Interventions: Drug: Placebo
- Reference Drug (Active Comparator): Cetirizine
  Interventions: Drug: Cetirizine

INTERVENTIONS:
Drug: ACT-129968 — daily tablets
  Other Names: Setipiprant
  Arms: Investigational Drug
Drug: Placebo — matching placebo tablets and capsules
  Arms: Comparative Drug
Drug: Cetirizine — daily capsules
  Arms: Reference Drug

SUMMARY:
This study will assess the efficacy and safety of ACT-129968 in adolescent, adult and elderly patients with seasonal allergic rhinitis, due to mountain cedar pollen.

ELIGIBILITY:
Inclusion Criteria

* Males and females aged 12-76 years with documented clinical history of symptomatic seasonal allergic rhinitis associated with mountain cedar pollen for the last 2 years.
* Evening reflective Total Nasal Symptom Score (p.m.rTNSS) at least 42 out of a maximum potential score of 84 over the 7-day run-in period, or > or = 6 out of a maximum score of 12 on each of the last 4 consecutive days during the run-in period.

Exclusion Criteria

* Non-allergic rhinitis.
* Severe physical nasal obstruction.
* Acute or significant chronic sinusitis.
* Bacterial or viral infection of the upper or lower respiratory tract, nasal sinuses, or middle ear.
* Ongoing chronic respiratory disorders.
* Asthma requiring use of short-acting beta2-agonists > 2 times a week or any asthma treatment other than inhaled short-acting beta2-agonists.
* Diagnosis of aspirin or non-steroidal anti-inflammatory drug (NSAID)-induced asthma.
* Nasal biopsy or surgery, sinus surgery, or perforation within the 8 weeks prior to the Screening Visit.
* Ocular surgery within the 8 weeks prior to the Screening Visit.
* Ocular infections (bacterial or viral) within the 4 weeks before screening.
* Use of forbidden medications (prescribed or over-the-counter [OTC])
* Congenital or acquired severe immunodeficiency or known Human immunodeficiency virus (HIV)infection.

Ages: 12 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The mean change in Daytime Nasal Symptom Score | baseline to end of treatment period (2 weeks)

SECONDARY OUTCOMES:
The mean change in other daytime/nighttime symptom scores of allergic rhinitis | baseline to end of treatment period (2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grabo, PhD, Study Director — Actelion
Locations (7):
- United States (7):
  - Clinical Investigative Site 7905, Austin, Texas
  - Clinical Investigative Site 7907, Kerrville, Texas
  - Clinical Investigative Site 7903, New Braunfels, Texas
  - Clinical Investigative Site 7901, San Antonio, Texas
  - Clinical Investigative Site 7902, San Antonio, Texas
  - Clinical Investigative Site 7904, San Antonio, Texas
  - Clinical Investigative Site 7906, San Antonio, Texas

REFERENCES:
- [Derived] Ratner P, Andrews CP, Hampel FC, Martin B, Mohar DE, Bourrelly D, Danaietash P, Mangialaio S, Dingemanse J, Hmissi A, van Bavel J. Efficacy and safety of setipiprant in seasonal allergic rhinitis: results from Phase 2 and Phase 3 randomized, double-blind, placebo- and active-referenced studies. Allergy Asthma Clin Immunol. 2017 Apr 4;13:18. doi: 10.1186/s13223-017-0183-z. eCollection 2017. PMID 28392807